CLINICAL TRIAL: NCT00450632
Title: CONSTITUTION D'UNE BIOTHEQUE DE PATIENTS DE SEINE-MARITIME AUX ANTECEDENTS D'INFECTION INVASIVE A MENINGOCOQUES
Brief Title: Creation of a Biotheque of Patients of Seine-Maritime With Meningococcal Infection
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2005/031/HP
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Meningococcal Infections
Keywords: meningococcal infections; biotheque; genetic markers
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main objective of this study is to constitute a biotheque of patients with meningococcal disease to enable results to be interpreted and genetic factors to be determined

ELIGIBILITY:
Inclusion Criteria:

* Subjects of Seine-Maritime with a meningococcal disease from the year of 2000
* parental authority assent if necessary

Exclusion Criteria:

* no parental authority assent
* child under supervision

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects of Seine-Maritime with a meningococcal disease
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2005-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: François Caron, Professor, Principal Investigator — University Hopital of Rouen
Locations (1):
- UH Rouen, Rouen, Seine-Maritime, France